CLINICAL TRIAL: NCT03486977
Title: Effectiveness and Organizational Conditions of Effectiveness of Telemedicine in Establishments Providing Care for the Dependent Elderly
Acronym: EFFORT
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2016/32
Record Dates: First submitted 2018-01-23; First posted 2018-04-03 (Actual); Last update posted 2020-01-07 (Actual); Status verified 2020-01

CONDITIONS: Health Services for the Aged
MeSH Terms: interventions — Telemedicine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Establishments with telemedicine system: Establishments equipped for telemedicine (teleconsultation, casualty) as part of the regional project of the Aquitaine regional program telemedicine device deployment.
  Interventions: Procedure: Evaluation of disease and follow-up
- Establishments without telemedicine system: Defined and equipped for telemedicine EHPAD after mating on the number of residents, the GMP (average weighted GIR), the PMP (weighted average PATHOS), the distance to a hospital with an emergency shelter service.
  The rate of unscheduled hospitalizations will be collected during follow-up visits in clinical departments of the healthcare of the Gironde by a research staff
  Interventions: Procedure: Evaluation of disease and follow-up

INTERVENTIONS:
Procedure: Evaluation of disease and follow-up — Correspondence medical consultation with specific device
  Other Names: Telemedicine

SUMMARY:
Study of interest of Telemedicine in establishments providing care for the dependent elderly (EHPAD in french) is a strategy for improving the course of care of residents, including the number not programmed hospitalizations, and a multidimensional analysis of the conditions of effectiveness of telemedicine will identify the keys to optimize its use.

DETAILED DESCRIPTION:
The project combines quantitative and qualitative analyses :

1. Quantitative study

Study of comparative prospective cohort clustered in two parallel groups:

Group 'Telemedicine': establishments providing care for the dependent elderly (EHPAD in french) equipped for telemedicine (teleconsultation, casualty) as part of the regional project of the Aquitaine Regional Agency of Heath telemedicine device deployment.

Control group: Defined and equipped for telemedicine EHPAD after matching on the number of residents, the GMP (average weighted GIR : "Groupes Iso Ressources" = score to reflects the average level of dependency of residents of a residential care facility for the elderly), the PMP (weighted average PATHOS = an evaluation system set up by the National Union of Clinical Gerontology and the Medical Service of the National Fund for Health Insurance for Salaried Workers), the distance to a hospital with an emergency shelter service.

The rate of unscheduled hospitalizations will be collected during follow-up visits in clinical departments of the healthcare of the Gironde (french department) by a research staff.

2 Qualitative study In the Group of nursing homes with telemedicine, said group "Telemedicine", will be identified four long-term care facilities, selected according to their degree of use of telemedicine (ratio number of teleconsultation per month / number of beds) (EHPAD 2 strong users, 2 nursing homes) low users) within these four long-term care facilities will be carried out observations of field and in-depth interviews with professionals, managers and attending physicians.

ELIGIBILITY:
Inclusion Criteria:

Quantitative research:

* All residents of nursing home men and women 65 years of age and more and likely to be eligible for a teleconsultation or a casualty because achieved one of the identified chronic pathologies as a reason for teleconsultation, will be included in both groups of long-term care
* Medical professionals working in the nursing home agreeing to answer the specifics questionnaires

Qualitative study:

* Doctors, physicians and coordinators nurses of Establishments Providing Care for the Dependent Elderly, nurses, orderly, psychologists, directors of Establishments
* Having a professional activity in nursing homes selected
* Having given their consent to participate in the study

Exclusion Criteria:

* Residents of long-term care facilities (quantitative study) Resident (or guardian/person) who expressed his opposition to participate in the study or not likely to be eligible for a teleconsultation or casualty Establishments Providing Care for the Dependent Elderly (qualitative) professionals
* Professional who expressed his opposition to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: All residents of EHPAD, men and women 65 years of age and more and likely to be eligible for a teleconsultation as suffering from one of the identified chronic pathologies as a reason for teleconsultation by Regional Agency of Hearth, will be included in the study in two groups of long-term care facilities. Eligible residents will be included in a very short time of 3 months.
Sampling Method: Probability Sample
Enrollment: 373 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-07-12 (Actual); Study Completion 2019-07-12 (Actual)

PRIMARY OUTCOMES:
Number of hospitalization not programmed residents on Medicine Surgery obstetrics (MCO) | 12 months
  Number of hospitalizations not programmed residents on Medicine Surgery obstetrics (MCO) between the inclusion and 12 month

SECONDARY OUTCOMES:
the main diagnosis, coded by the International Classification of diseases for every hospitalization | 12 months
  Evaluate the number of inappropriate hospitalization. The inappropriate hospitalization will be performed using the classification of Weissman. Weissman classification identifies causes of potentially preventable hospitalizations, from the main diagnosis, coded by the International Classification of diseases, version 10 (ICD10).
Score of the specific questionnaire for measurement of the context organizational and Managerial in health care facilities | 12 months
  Evaluate the impact of a strategy issued in EHPAD type teleconsultation or casualty on the quality of work life

CONTACTS AND LOCATIONS:
Overall Officials: Nathalie SALLES, MD, PhD, Principal Investigator — University Hospital, Bordeaux; Florence SALLIOUR, PhD, Study Chair — University Hospital, Bordeaux
Locations (24):
- France (24):
  - EHPAD CHU Bordeaux, Pessac, Lormont
  - EHPAD Le home medocain Arsac, Arsac
  - EHPAD Le parc du Bequet, Bègles
  - EHPAD Manon Cormier, Bègles
  - EHPAD Henry Dunant, Bordeaux
  - EHPAD Le Clos Serena, Bordeaux
  - EHPAD Résidence les Carmes, Bordeaux
  - EHPAD Cos villa Pia, Bordeaux
  - EHPAD Grand Bon Pasteur, Bordeaux
  - EHPAD Residence Aime Cesaire, Bordeaux
  - EHPAD Le Platane du Grand Parc, Bordeaux
  - EHPAD Seguin, Cestas
  - EHPAD résidence du Tertre, Fronsac
  - EHPAD Douceur de France, Gradignan
  - EHPAD Résidence l'Arousiney, Gujan-Mestras
  - EHPAD Le rétou, Lamarque
  - EHPAD Les coteaux, Lormont
  - Résidence de Médicis, Mérignac
  - EHPAD Fontaudin, Pessac
  - EHPAD Villa presentine, Rauzan
  - EHPAD Jacqueline Auriol, Saint-Seurin-sur-l'Isle
  - EHPAD Résidence La berge du lac, Talence
  - EHPAD Villa Bontemps, Talence
  - EHPAD Home Marie Curie, Villenave-d'Ornon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Han JH, Morandi A, Ely EW, Callison C, Zhou C, Storrow AB, Dittus RS, Habermann R, Schnelle J. Delirium in the nursing home patients seen in the emergency department. J Am Geriatr Soc. 2009 May;57(5):889-94. doi: 10.1111/j.1532-5415.2009.02219.x. PMID 19484845
- [Result] Morandi A, Han JH, Callison C, Ely EW, Schnelle JF. Delirium in nursing home residents across care transitions: a preliminary report. J Am Geriatr Soc. 2009 Oct;57(10):1956-8. doi: 10.1111/j.1532-5415.2009.02472.x. No abstract available. PMID 19807810
- [Result] Vellas B. Integrating Frailty into Clinical Practice to Prevent the Risk of Dependency in the Elderly. Nestle Nutr Inst Workshop Ser. 2015;83:99-104. doi: 10.1159/000382092. Epub 2015 Oct 20. PMID 26485153
- [Result] Graverholt B, Forsetlund L, Jamtvedt G. Reducing hospital admissions from nursing homes: a systematic review. BMC Health Serv Res. 2014 Jan 24;14:36. doi: 10.1186/1472-6963-14-36. PMID 24456561
- [Derived] Salles N, Saillour-Glenisson F, Sibe M, Langlois E, Kret M, Durrieu J, Arditi N, Abraham M, Perry F. Effectiveness and organizational conditions of effectiveness of telemedicine in nursing homes. A study protocol of a comparative prospective cohort (EFFORT study). Digit Health. 2021 Jan 24;7:2055207620982422. doi: 10.1177/2055207620982422. eCollection 2021 Jan-Dec. PMID 33598307